CLINICAL TRIAL: NCT04350125
Title: A Pilot Study Evaluating the Use of Autologous Platelet-rich Plasma (PRP) for the Treatment of Erectile Dysfunction
Brief Title: PRP for the Treatment of Erectile Dysfunction (ED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Gregory A. Broderick, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 18-010364
Record Dates: First submitted 2020-04-14; First posted 2020-04-16 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Intervention Model Description: Subjects treated in this study will be divided into 3 cohorts of 5. After the first cohort of 5 subjects have been treated and evaluated for safety, the second cohort of 5 subjects will proceed with treatment followed by review of events for safety. If determined safe to proceed the third cohort of 5 subjects will proceed with treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Platelet Rich Plasma Treatment (Experimental): Male subjects diagnosed with Erectile Dysfunction (ED) will receive platelet rich plasma injections.
  Interventions: Biological: Autologous Platelet Rich Plasma

INTERVENTIONS:
Biological: Autologous Platelet Rich Plasma — One 4-5mL platelet rich plasma injection administered to each side of the intracavernosal space on the right and left side of the corpus cavernosum at the base of the penis, every two weeks for 6 weeks.

SUMMARY:
Researchers are trying to determine the safety and efficacy of Platelet Rich Plasma (PRP) in the treatment of Erectile Dysfunction (ED).

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his informed and signed written consent
* The patient has ED for longer than 1 year but less than 5 years.
* The subject has a stable partner for at least 3 months.
* The patient is PDE5i responsive, meaning he is able to achieve and maintain an erection under the effect of the maximal dosage of PDE5i
* IIEF-EF, EHS, SEP 2+3, and GAQ Domain score of 17-20 Mild to moderate vascular erectile dysfunction: PSV > 25 cm/sec

Exclusion Criteria:

The patient is participating in another study that may interfere with the results or conclusions of this study

* History of radical prostatectomy or pelvic cancer surgery
* Prior history of pelvic malignancies
* Prior pelvic radiation therapy
* Neurological disease which effects erectile function (Spinal cord injury, iatrogenic injury to the pelvic or cavernous nerves)
* Psychiatric disease which effects erectile function
* The patient is taking blood thinners
* History of Diabetes Mellitus
* History of Coronary Artery Disease
* Evidence Based Criteria: Doppler Clinical Exam ( PSV < 25 cm/sec defined criteria for severe erectile dysfunction not likely to respond to approved medical therapies)
* Biochemical evidence of Hypogonadism (total Testosterone < 300 ng/dL)

Ages: 45 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-03-04 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-10-23 (Actual)

PRIMARY OUTCOMES:
Treatment-related adverse events | 35 weeks
  Number of participants to experience treatment-related adverse events defined as reaction in the skin (e.g., swelling, erythema, and warmth), injection site discomfort, penile pain, change in penile appearance, novel sexual concerns and any systemic reactions seen by the investigators, or concerns expressed by patients.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Broderick, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials